CLINICAL TRIAL: NCT04447326
Title: Randomized Controlled, Multicenter Phase II Clinical Research of Toripalimab (PD-1 Inhibitor) and Endostar Combined With Radiotherapy and Chemotherapy in the Treatment of High-risk Locally Advanced Nasopharyngeal Carcinoma
Brief Title: Toripalimab, Endostar Combined With Radiotherapy and Chemotherapy for Nasopharyngeal Carcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: First Affiliated Hospital of Guangxi Medical University (Other)
Collaborators: Shandong Cancer Hospital and Institute (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); The Affiliated Hospital Of Guizhou Medical University (Other); Xiangya Hospital of Central South University (Other); Jiangxi Provincial Cancer Hospital (Other); Zhejiang Cancer Hospital (Other); Fourth Affiliated Hospital of Guangxi Medical University (Other); LiuZhou People's Hospital (Other); Guilin Medical College (Other); Afﬁliated Hospital of North Sichuan Medical College (Other)
Responsible Party: Principal Investigator, min kang, professor, First Affiliated Hospital of Guangxi Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FirstGuangxiMU1
Record Dates: First submitted 2020-06-23; First posted 2020-06-25 (Actual); Last update posted 2020-06-25 (Actual); Status verified 2020-06

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — toripalimab; Radiotherapy; Drug Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- IC＋CCRT＋Toripalimab＋Endostar (Experimental): Three cycles of induction chemotherapy with GP regimen (Q3W): Gem 1000 mg/m2 d1,8; DDP 80mg/m2 d1, Q3W; IMRT (6-7 weeks, 5 times each week) combined with cisplatin for 2-3 cycles (Q3W): DDP 100 mg/m2, Q3W, 2-3 cycles; IMRT: GTVnx 70-74Gy/30-33f, 5d/w, 6-7 w; Toripalimab: 240 mg, Q3W, starting on D1, for totally 12 cycles; Endostar: 7.5 mg/m2/d, continuous intravenous pumping for 10 days, Q3W, starting on D1, for totally 5 cycles.
  Interventions: Drug: Toripalimab, Endostar Combined With Radiotherapy and Chemotherapy
- IC＋CCRT (Active Comparator): Three cycles of induction chemotherapy with GP regimen (Q3W): Gem 1000 mg/m2 d1,8; DDP 80mg/m2 d1, Q3W; IMRT (6-7 weeks, 5 times each week) combined with cisplatin for 2-3 cycles (Q3W): DDP 100 mg/m2, Q3W, 2-3 cycles; IMRT: GTVnx 70-74Gy/30-33f, 5d/w, 6-7 w.
  Interventions: Drug: IC＋CCRT

INTERVENTIONS:
Drug: Toripalimab, Endostar Combined With Radiotherapy and Chemotherapy — Toripalimab: 240 mg, Q3W, starting on D1, for totally 12 cycles Endostar: 7.5 mg/m2/d, continuous intravenous pumping for 10 days, Q3W, starting on D1, for totally 5 cycles
  Other Names: JS001
  Arms: IC＋CCRT＋Toripalimab＋Endostar
Drug: IC＋CCRT — IC＋CCRT
  Arms: IC＋CCRT

SUMMARY:
This study is to investigate the efficacy and safety of the induction chemotherapy + concurrent chemoradiotherapy（CCRT）combined with toripalimab and endostar treatment, in comparison with the induction chemotherapy + concurrent chemoradiotherapy（CCRT）, in treating locally advanced high-risk nasopharyngeal carcinoma

DETAILED DESCRIPTION:
GP-induced chemotherapy combined with concurrent chemoradiotherapy is the standard treatment for the locally advanced nasopharyngeal carcinoma recommended by the guidelines. However, the prognosis for T4 and/or N3 nasopharyngeal carcinoma is still poor, with the 3-year PFS of about 70%. Therefore, it is of great importance to improve the prognosis of patients with locally advanced high-risk nasopharyngeal carcinoma. Immunotherapy has been an emerging treatment method for tumors in recent years. Compared with the chemotherapy, immunotherapy has less adverse reactions, and the effects could last longer, significantly improving the prognosis and patients' quality of life. Endostar, as a VEGFR inhibitor, has good safety in treating nasopharyngeal carcinoma. Related data have shown that PD-1 and Endostar exert synergistic antitumor effects in a mouse model of lung cancer. A Phase II multi-center clinical study from our center has shown that, for patients with locally advanced low-risk nasopharyngeal carcinoma, all the 3-year OS, PFS, and DMFS for the radiotherapy combined with Endostar group were superior to the concurrent chemoradiotherapy group, and the combination of radiotherapy and Endostar lead to significantly reduced adverse effects. In clinical studies concerning other solid tumors, it has also been observed that the PD-1 inhibitors combined with VEGFR inhibitors could significantly improve the efficacy, and achieve synergistic effects. Therefore, A Phase II，randomized, prospective, multicentric clinical trail was conducted to compare the efficacy and safety of induction chemotherapy and the concurrent chemoradiotherapy plus Endostar and PD-1, followed by PD-1 treatment for half a year compared with the induction chemotherapy and the concurrent chemoradiotherapy for the T4 and/or N3 nasopharyngeal carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. With ECOG score 0-1.
2. Subjective aged 18-65 years, male or non-pregnant female.
3. Pathologically diagnosed as nasopharyngeal non-keratinizing carcinoma (differentiated or undifferentiated, i.e., the WHO type II or III).
4. Stage IVa (8th AJCC/UICC stage) T4 and/or N3, untreated patients with nasopharyngeal carcinoma.
5. Agreeing to provide previously stored tumor tissue samples or perform biopsy to collect tumor tissues, which were sent to the central laboratory for the PD-L1 IHC test.
6. Hematology: white blood cells ≥ 4000 /μL; neutrophils ≥ 2000 /μL; hemoglobin ≥ 9 g/dL; and platelets ≥ 100000 /μL.
7. Liver function: ALT and AST lower than the 1.5 times (1.5 × ) the upper limits of normal (ULN); and total bilirubin < 1.5 × ULN.
8. Renal function: serum creatinine < 1.5 × ULN.
9. Patients signing the informed consents, and willing and able to follow the study plan (visit and treatment plan), laboratory tests, and other research procedures.

Exclusion criteria:

1. Patients with nasopharyngeal carcinoma with recurrence and distant metastasis.
2. Pathologically diagnosed as keratinizing squamous cell carcinoma (WHO classification type I).
3. Patients who had undergone radiotherapy or systemic chemotherapy.
4. Pregnant or breastfeeding females, or females in fertility period while with no effective contraceptive measures.
5. Positive for HIV.
6. Having suffered from other malignant tumors (except for the cured basal cell carcinoma or cervical carcinoma in situ).
7. Having been treated with inhibitors of immune regulatory points (i.e., CTLA-4, PD-1, PD-L1, etc.).
8. With complications needing long-term application of immunosuppressive drugs, or systemic or local application of corticosteroids with immunosuppressive doses of comorbidities.
9. Patients with immunodeficiency diseases, or a history of organ transplantation (including but not limited to: interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary inflammation, nephritis, hyperthyroidism, hypothyroidism; patients suffering from vitiligo, or asthma in childhood completely relieved, with no need of any intervention after adulthood could be included; and patients with asthma requiring bronchodilators for medical intervention could not be included).
10. With excessive usage of glucocorticoids within 4 weeks.
11. Whose laboratory examination values that did not meet the relevant standards within 7 days before participating in the research.
12. Patients with markedly reduced heart, liver, lung, kidney and/or bone marrow functions.
13. With serious and uncontrolled medical diseases and infections.
14. Using other test drugs or in other clinical trials.
15. Refusing or failing to sign the informed consent to participate in the trial.
16. With other treatment contraindications.
17. With personality or mental illness, with no or limited civil capacity.
18. Positive for hepatitis B surface antigen (HBsAg), and peripheral blood hepatitis B virus deoxyribonucleic acid (HBV DNA) ≥ 1000 cps/mL.
19. Patients positive for the HCV antibody test could only be included in this study with the negative results from the HCV RNA polymerase chain reaction test.
20. Unable to cooperate with regular follow-up due to psychological, social, family and geographical reasons.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2020-06 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
progression-free survival, PFS | 3 years
  calculated from the date of randomisation to the date of the documented local or regional relapse, distant metastasis, or death from any cause, whichever occurred first. distant failure, or death from any cause, whichever occurred first.

SECONDARY OUTCOMES:
Overall Survival，OS | 3 years
  the time from random assignment to death from any cause or censored at the date of last follow-up.
locoregional relapse-free Survival, LRFS | 3 years
  the time from random assignment to local or regional relapse.
Distant metastasis-free survival,DMFS | 3 years
  calculated from date of randomisation to the first distant failure
Overall response rate (ORR) | 3 months
  complete response (CR) + partial response (PR)
adverse events (AEs) and severe adverse events (SAE) | 3 years
  graded according to NCI CTCAE 5.0

REFERENCES:
- [Background] Zhang S, Huang X, Zhou L, Wu G, Lin J, Yang S, Chen J, Lin S. An open-label, single-arm phase II clinical study of induction chemotherapy and sequential Nimotuzumab combined with concurrent chemoradiotherapy in N3M0 stage nasopharyngeal carcinoma. J BUON. 2018 Nov-Dec;23(6):1656-1661. PMID 30610791
- [Background] Hsu C, Lee SH, Ejadi S, Even C, Cohen RB, Le Tourneau C, Mehnert JM, Algazi A, van Brummelen EMJ, Saraf S, Thanigaimani P, Cheng JD, Hansen AR. Safety and Antitumor Activity of Pembrolizumab in Patients With Programmed Death-Ligand 1-Positive Nasopharyngeal Carcinoma: Results of the KEYNOTE-028 Study. J Clin Oncol. 2017 Dec 20;35(36):4050-4056. doi: 10.1200/JCO.2017.73.3675. Epub 2017 Aug 24. PMID 28837405
- [Background] Ma BBY, Lim WT, Goh BC, Hui EP, Lo KW, Pettinger A, Foster NR, Riess JW, Agulnik M, Chang AYC, Chopra A, Kish JA, Chung CH, Adkins DR, Cullen KJ, Gitlitz BJ, Lim DW, To KF, Chan KCA, Lo YMD, King AD, Erlichman C, Yin J, Costello BA, Chan ATC. Antitumor Activity of Nivolumab in Recurrent and Metastatic Nasopharyngeal Carcinoma: An International, Multicenter Study of the Mayo Clinic Phase 2 Consortium (NCI-9742). J Clin Oncol. 2018 May 10;36(14):1412-1418. doi: 10.1200/JCO.2017.77.0388. Epub 2018 Mar 27. PMID 29584545
- [Background] Li Y, Tian Y, Jin F, Wu W, Long J, Ouyang J, Zhou Y. A phase II multicenter randomized controlled trial to compare standard chemoradiation with or without recombinant human endostatin injection (Endostar) therapy for the treatment of locally advanced nasopharyngeal carcinoma: Long-term outcomes update. Curr Probl Cancer. 2020 Feb;44(1):100492. doi: 10.1016/j.currproblcancer.2019.06.007. Epub 2019 Jul 2. PMID 32035692
- [Background] Kang M, Wang F, Liao X, Zhou P, Wang R. Intensity-modulated radiotherapy combined with endostar has similar efficacy but weaker acute adverse reactions than IMRT combined with chemotherapy in the treatment of locally advanced nasopharyngeal carcinoma. Medicine (Baltimore). 2018 Jun;97(25):e11118. doi: 10.1097/MD.0000000000011118. PMID 29924009